CLINICAL TRIAL: NCT00699959
Title: Comparison and Description of Coronary Patients Management With or Without Heart Failure in Cardiology Consulting
Brief Title: National Survey on Coronary Patients and Heart Failure Performed in 2 Patient Groups
Acronym: COMPAR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2007/8
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Patients; Heart Failure
Keywords: Coronary patients; heart failure; dyslipidemia
MeSH Terms: conditions — Heart Failure; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with heart failure
- 2: patients without heart failure

SUMMARY:
The purpose of this observational study is to compare frequency of attainment control goals through the more represented cardiovascular factor risk, dyslipidemia, among coronary patients with or without heart failure in cardiology consulting.

ELIGIBILITY:
Inclusion Criteria:

* patient with coronary disease diagnosed since at least 1 year
* Echocardiography done less than 1 year ago
* patient with or without documented heart failure

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First two consecutive Coronary patients with or without heart failure
Sampling Method: Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2008-06; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of attainment control goals through the more represented cardiovascular factor risk, dyslipidemia, among coronary patients with or without heart failure in cardiology consulting. | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Study Director — AstraZeneca
Locations (324):
- France (324):
  - Research Site, Abbeville
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Amboise
  - Research Site, Amiens
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annemasse
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Arès
  - Research Site, Argentan
  - Research Site, Arles
  - Research Site, Armentières
  - Research Site, Arnouville
  - Research Site, Arras
  - Research Site, Asnières-sur-Seine
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Audincourt
  - Research Site, Aulnay-sous-Bois
  - Research Site, Avallon
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bagnolet
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Bailleul
  - Research Site, Balma
  - Research Site, Bar-le-Duc
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Beaumont-de-Lomagne
  - Research Site, Beausoleil
  - Research Site, Beauvais
  - Research Site, Belfort
  - Research Site, Belley
  - Research Site, Bergerac
  - Research Site, Besançon
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Blois
  - Research Site, Bois-Colombes
  - Research Site, Bois-Guillaume
  - Research Site, Bonneuil-sur-Marne
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourges
  - Research Site, Brest
  - Research Site, Briey
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cahors
  - Research Site, Cannes
  - Research Site, Cannes La Bocca
  - Research Site, Carcassonne
  - Research Site, Carpentras
  - Research Site, Castelnaudary
  - Research Site, Castres
  - Research Site, Cavaillon
  - Research Site, Cenon
  - Research Site, Cergy
  - Research Site, Cesson-Sévigné
  - Research Site, Challans
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Chamonix
  - Research Site, Champigny-sur-Marne
  - Research Site, Chantilly
  - Research Site, Charleville-Mézières
  - Research Site, Chartres
  - Research Site, Chaville
  - Research Site, Château-d'Olonne
  - Research Site, Châteaubernard
  - Research Site, Châteauroux
  - Research Site, Châtillon
  - Research Site, Châtillon-sur-Seine
  - Research Site, Cherbourg Octeville
  - Research Site, Choisy-le-Roi
  - Research Site, Cholet
  - Research Site, Clamart
  - Research Site, Clermont-Ferrand
  - Research Site, Commercy
  - Research Site, Condé-sur-l'Escaut
  - Research Site, Conflans STE Honorine
  - Research Site, Corbeil-Essonnes
  - Research Site, Cornebarrieu
  - Research Site, Cournon-d'Auvergne
  - Research Site, Coutances
  - Research Site, Creil
  - Research Site, Croix
  - Research Site, Dax
  - Research Site, Denain
  - Research Site, Décines-Charpieu
  - Research Site, Dieulefit
  - Research Site, Dijon
  - Research Site, Divion
  - Research Site, Dol-de-Bretagne
  - Research Site, Douai
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Dunkirk
  - Research Site, Erstein
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Étampes
  - Research Site, Évecquemont
  - Research Site, Évian-les-Bains
  - Research Site, Floirac
  - Research Site, Frontignan
  - Research Site, Genas
  - Research Site, Gennevilliers
  - Research Site, Grande-Synthe
  - Research Site, Grenoble
  - Research Site, Grésy-sur-Aix
  - Research Site, Guebwiller
  - Research Site, Guéret
  - Research Site, Guyancourt
  - Research Site, Haguenau
  - Research Site, Harfleur
  - Research Site, Hayange
  - Research Site, Hazebrouck
  - Research Site, Hesdin
  - Research Site, Hénin-Beaumont
  - Research Site, Hyères
  - Research Site, Issy-les-Moulineaux
  - Research Site, Juan-les-Pins
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Île-Rousse
  - Research Site, La Bassée
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, La Ciotat
  - Research Site, La Courneuve
  - Research Site, La Flèche
  - Research Site, La Madeleine
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Verpillière
  - Research Site, Lagny-sur-Marne
  - Research Site, Lamballe
  - Research Site, Lanester
  - Research Site, Langon
  - Research Site, Lannemezan
  - Research Site, Le Bourget
  - Research Site, Le Chesnay
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Port-Marly
  - Research Site, Le Raincy
  - Research Site, Les Clayes-sous-Bois
  - Research Site, Les Sables-d'Olonne
  - Research Site, Les Ulis
  - Research Site, Levallois-Perret
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Limoux
  - Research Site, Lisieux
  - Research Site, Lomme
  - Research Site, Longeville-lès-Metz
  - Research Site, Lons-le-Saunier
  - Research Site, Lorient
  - Research Site, Lunel
  - Research Site, Lyon
  - Research Site, Malo-les-Bains
  - Research Site, Marcq-en-Barœul
  - Research Site, Marcy-l'Étoile
  - Research Site, Maromme
  - Research Site, Marseille
  - Research Site, Maubeuge
  - Research Site, Maurepas
  - Research Site, Mayenne
  - Research Site, Mâcon
  - Research Site, Meaux
  - Research Site, Mende
  - Research Site, Menton
  - Research Site, Metz
  - Research Site, Millau
  - Research Site, Milly-la-Forêt
  - Research Site, Miramas
  - Research Site, Monaco
  - Research Site, Mont-de-Marsan
  - Research Site, Montargis
  - Research Site, Montauban
  - Research Site, Montesson
  - Research Site, Montélimar
  - Research Site, Montfermeil
  - Research Site, Montigny-lès-Metz
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Morlaix
  - Research Site, Mulhouse
  - Research Site, Muret
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Neufchâteau
  - Research Site, Neuville-sur-Saône
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Noisy-le-Grand
  - Research Site, Olivet
  - Research Site, Ollioules
  - Research Site, Orléans
  - Research Site, Ornans
  - Research Site, Orsay
  - Research Site, Oullins
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Palaiseau
  - Research Site, Pantin
  - Research Site, Paray-le-Monial
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Périgueux
  - Research Site, Pithiviers
  - Research Site, Plaisance-du-Touch
  - Research Site, Plan-de-Cuques
  - Research Site, Ploërmel
  - Research Site, Poitiers
  - Research Site, Pont-à-Mousson
  - Research Site, Pontarlier
  - Research Site, Pontault-Combault
  - Research Site, Pontoise
  - Research Site, Prévessin-Moëns
  - Research Site, Quimper
  - Research Site, Quincy-sous-Sénart
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Revel
  - Research Site, Ris-Orangis
  - Research Site, Rodez
  - Research Site, Rognac
  - Research Site, Romans-sur-Isère
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Royat
  - Research Site, Rueil-Malmaison
  - Research Site, Sablé-sur-Sarthe
  - Research Site, Saint-Avertin
  - Research Site, Saint-Avold
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Chamond
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Etienne
  - Research Site, Saint-Fargeau-Ponthierry
  - Research Site, Saint-Fons
  - Research Site, Saint-Genis-Laval
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Gély-du-Fesc
  - Research Site, Saint-Julien-en-Genevois
  - Research Site, Saint-Louis
  - Research Site, Saint-Lô
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Ouen
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pol-de-Léon
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Raphaël
  - Research Site, Sanary-sur-Mer
  - Research Site, Sarcelles
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sceaux
  - Research Site, Schiltigheim
  - Research Site, Sélestat
  - Research Site, Somain
  - Research Site, Sorgues
  - Research Site, St.-Jean
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Tarbes
  - Research Site, Taverny
  - Research Site, Tergnier
  - Research Site, Ternay
  - Research Site, Thann
  - Research Site, Thiais
  - Research Site, Thionville
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tournefeuille
  - Research Site, Tours
  - Research Site, Trappes
  - Research Site, Troyes
  - Research Site, Ussel
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Vannes
  - Research Site, Vernon
  - Research Site, Vernouillet
  - Research Site, Vesoul
  - Research Site, Vénissieux
  - Research Site, Villecresnes
  - Research Site, Villefranche-de-Lauragais
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villejuif
  - Research Site, Villeneuve Saint Georges CEDE
  - Research Site, Villeneuve-le-Roi
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villeparisis
  - Research Site, Villepreux
  - Research Site, Villeurbanne
  - Research Site, Vincennes
  - Research Site, Viroflay
  - Research Site, Vitré
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittel
  - Research Site, Wattrelos